CLINICAL TRIAL: NCT04758260
Title: Influence of the Antioxidant Treatment in the Oxidant-reduction Potential in Seminal Plasma in Men Whose Partners Will Undergo Through an Egg Donation Cycle
Acronym: Mioxsys ox
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty recruiting
Sponsor: IVI Bilbao (Other)
Collaborators: Aytu BioPharma, Inc. (Industry)
Responsible Party: Principal Investigator, FERNANDO QUINTANA FERRAZ, Marcos Ferrando Serrano, IVI Bilbao
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1708-BIO-088-MM
Record Dates: First submitted 2020-03-09; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Compare the sORP Rate in Sperm Samples, Obtained by the Mioxsys System, Before and After 2.5 Months Antioxidant Men Supplements Treatment (Fertybiotic Man)
MeSH Terms: interventions — Antioxidants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Antioxidant Treatment (Experimental): Influence of the Antioxidant Treatment in the Oxidant-reduction Potential in Seminal Plasma in Men
  Interventions: Dietary Supplement: Antioxidant

INTERVENTIONS:
Dietary Supplement: Antioxidant — Oral antioxidant oral intake in the 3 months prior to inclusion in the study

SUMMARY:
Evaluate the influence of antioxidant men supplements treatment (Fertybiotic Hombre) in the rate of sORP (stactic Oxidation Reduction Potential) defined as the balanced measure between the total oxidant activity (ROS, superoxides, nitric oxide, peroxide) and total reducing activity (alpha tocopherol, β carotene, uric acid) in sperm samples during egg donation cycles.

We will also evaluate the influence of the sORP rate in the embryo development during the egg donation treatments; taking in account the fecundation rate, percentage of blastocyst stage arrival embryos, number of frozen embryos, implantation rate, on-going pregnancy rate and miscarriage rate.

The sperm sample will be measured by electrochemical technology using Mioxsys system for a quantitative measurement in millivolts (mV), in those male patients who participate in an egg donation assisted reproduction treatment.

After 14 days, the pregnancy stage will be available. This information will be obtained from the patient's clinical history using the human chorionic gonadotropin hormone (shCG) in blood. It will be performed either in our Clinic or externally within the usual practice derived from the treatment carried out. These values will be compared with the results obtained from sORP.

ELIGIBILITY:
Male Inclusion Criteria

* Sperm count greater than 2 million per milliliter
* Sperm origin: ejaculate

Exclusion Criteria:

* Taking oral antioxidants in the 3 months prior to inclusion in the study
* Total astenozoospermia or Severe teratozoospermia (including balloonzoospermia)

Ages: 18 Years to 48 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2021-02-12 (Actual)

PRIMARY OUTCOMES:
Compare the sORP rate in sperm samples, | 2.5 months
  Compare the sORP rate in sperm samples, obtained by the Mioxsys System, before and after 2.5 months antioxidant men supplements treatment (Fertybiotic MAN).

SECONDARY OUTCOMES:
Evaluate the influence of the sORP rate in embryo development | 1 year
  Analysis of different embryo quality parameters as:
  * fecundation rate
  * percentage of blastocyst stage arrival embryos
  * number of frozen embryos
Evaluate the relationship between the sORP rate in sperm samples | 1 year
  Evaluate the relationship between the sORP rate in sperm samples, obtained by Mioxsys System, with the implantation rate, on-going pregnancy rate and miscarriage rate.
Determinate a reproductive prognosis value based on sORP rate and the different sperm parameters | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marcos Ferrando, Principal Investigator — IVI Bilbao
Locations (1):
- IVI Bilbao, Leioa, Vizcaya, Spain

IPD SHARING:
Plan to Share IPD: No